CLINICAL TRIAL: NCT00614848
Title: Randomized Controlled Trial to Evaluate the Safety and Efficacy of the Medtronic AVE ABT-578 Eluting Driver Coronary Stent in De Novo Native Coronary Artery Lesions
Brief Title: The ENDEAVOR II Clinical Trial: The Medtronic Endeavor Drug Eluting Coronary Stent System in Coronary Artery Lesions
Acronym: ENDEAVOR II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Judith L. Jaeger, Director of Clinical Research, Medtronic Vascular
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IP034
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Coronary Artery Disease; Arterial Occlusive Diseases; Coronary Disease; Coronary Arteriosclerosis; Heart Diseases; Myocardial Ischemia; Vascular Diseases; Ischemia; Arteriosclerosis
Keywords: restenosis
MeSH Terms: conditions — Coronary Artery Disease; Arterial Occlusive Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia; Vascular Diseases; Ischemia; Arteriosclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Endeavor Drug Eluting Coronary Stent
  Interventions: Device: Endeavor drug eluting coronary stent
- 2 (Active Comparator): Driver bare-metal coronary stent
  Interventions: Device: Endeavor drug eluting coronary stent

INTERVENTIONS:
Device: Endeavor drug eluting coronary stent — Zotarolimus coated coronary stent (10ug/mm)

SUMMARY:
To demonstrate the safety and efficacy of the Driver Coronary Stent coated with 10 mcg/mm ABT-578 compared to the uncoated Driver Stent for the treatment of single de novo lesions in native coronary arteries 2.25-3.5 mm in diameter.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an acceptable candidate for PTCA, stenting, and emergent CABG.
* Subject must have clinical evidence of ischemic heart disease or a positive functional study.
* Subject has single vessel disease or has multivessel disease with only moderate stenosis (max 50-60% or total occlusion (100%) for which no interventions are planned at the time of study inclusion).
* Target lesion / vessel must meet the following criteria:

  1. Target lesion is a single de novo lesion that has not been previously treated with any interventional procedure. Only one lesion may be treated per subject
  2. Target vessel must be a native coronary artery with a stenosis of >=50% and <100%
  3. Target lesion must be >= 14 mm and ≤ 27 mm in length
  4. Target vessel reference diameter must be >= 2.25 mm and ≤3.5 mm
* Female subjects of childbearing potential must have a negative pregnancy test within 7 days before the procedure.
* Subject or subject's legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical site
* Subject and treating physician agree that subject will comply with all required post-procedure follow-up

Exclusion Criteria:

* A documented left ventricular ejection fraction <30%
* A known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, cobalt, nickel, chromium, or a sensitivity to contrast media, which cannot be adequately pre-medicated
* History of an allergic reaction or significant sensitivity or receiving drugs similar to/or synergistic to ABT-578 (rapamycin, tacrolimus, sirolimus, CCI-779 or other analogues).
* A platelet count <100,000 cells/mm³ or >700,000 cells/mm³, or a WBC <3,000 cells/mm³
* Evidence of an acute myocardial infarction within 72 hours of the intended treatment (defined as: Q wave or non-Q wave infarction having CK enzymes >2X the upper laboratory normal with the presence of a CK-MB elevated above the Institution's upper limit of normal).
* Creatinine >2.0 mg/dl
* A previous coronary interventional procedure of any kind within the 30 days prior to the procedure
* Subject requires planned interventional treatment of either the target or any non-target vessel within 30 days post-procedure
* Target lesion requires treatment with a device other than PTCA prior to stent placement
* Previous stenting anywhere in the target vessel
* Target vessel has evidence of thrombus or is excessively tortuous (2 bends >90 degrees to reach the target lesion)
* Significant (>50%) stenosis proximal or distal to the target lesion that might require revascularization or impede run off
* Target lesion located in native vessel distally to anastomosis with vein graft or LIMA
* Target lesion has any of the following characteristics:

  1. Lesion location is aorto-ostial, an unprotected left main lesion, or within 5mm of the origin of the LAD, LCX, or RCA
  2. Involves a side branch >2.0 mm in diameter
  3. Is at or distal to a 45º bend in the vessel
  4. Is severely calcified
* Unprotected left main coronary artery disease (an obstruction greater than 50% in the left main coronary artery)
* History of a stroke or transient ischemic attack within the prior 6 months
* Active peptic ulcer or upper GI bleeding within the prior 6 months
* The subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Concurrent medical condition with a life expectancy of less than 12 months
* Any previous or planned treatment with anti-restenotic therapies including, but not limited to, drug-eluting stents and brachytherapy
* Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2003-06; Primary Completion 2005-01 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure Rate at 9 months post procedure | 9 months

SECONDARY OUTCOMES:
Device Success Lesion Success Procedure Success Major Cardiac Adverse Events (MACE) at 30 days and 6, 9, and 12 months, and annually thereafter out to 5 years. Late loss at 8 months as measured by QCA | 30 days and 6, 9, and 12 months, and annually thereafter out to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: J. Fajadet, MD, Principal Investigator — Clinique Pasteur, France; Richard E Kuntz, MD, MSc, Principal Investigator — Harvard Medical School, USA; W. Wijns, MD, PhD, Principal Investigator — OLV Hospital, Belgium
Locations (1):
- Dr. J. Fajedet, Clinique Pasteur, France

REFERENCES:
- [Result] Fajadet J, Wijns W, Laarman GJ, Kuck KH, Ormiston J, Munzel T, Popma JJ, Fitzgerald PJ, Bonan R, Kuntz RE; ENDEAVOR II Investigators. Randomized, double-blind, multicenter study of the Endeavor zotarolimus-eluting phosphorylcholine-encapsulated stent for treatment of native coronary artery lesions: clinical and angiographic results of the ENDEAVOR II trial. Circulation. 2006 Aug 22;114(8):798-806. doi: 10.1161/CIRCULATIONAHA.105.591206. Epub 2006 Aug 14. PMID 16908773
- [Derived] Mauri L, Massaro JM, Jiang S, Meredith I, Wijns W, Fajadet J, Kandzari DE, Leon MB, Cutlip DE, Thompson KP. Long-term clinical outcomes with zotarolimus-eluting versus bare-metal coronary stents. JACC Cardiovasc Interv. 2010 Dec;3(12):1240-9. doi: 10.1016/j.jcin.2010.08.021. PMID 21232717
- [Derived] Remak E, Manson S, Hutton J, Brasseur P, Olivier E, Gershlick A. Cost-effectiveness of the Endeavor stent in de novo native coronary artery lesions updated with contemporary data. EuroIntervention. 2010 Feb;5(7):826-32. doi: 10.4244/eijv5i7a138. PMID 20142198
- [Derived] Eisenstein EL, Wijns W, Fajadet J, Mauri L, Edwards R, Cowper PA, Kong DF, Anstrom KJ. Long-term clinical and economic analysis of the Endeavor drug-eluting stent versus the Driver bare-metal stent: 4-year results from the ENDEAVOR II trial (Randomized Controlled Trial to Evaluate the Safety and Efficacy of the Medtronic AVE ABT-578 Eluting Driver Coronary Stent in De Novo Native Coronary Artery Lesions). JACC Cardiovasc Interv. 2009 Dec;2(12):1178-87. doi: 10.1016/j.jcin.2009.10.011. PMID 20129543